CLINICAL TRIAL: NCT05178290
Title: Back to ECE Safely With SAGE: Reducing COVID-19 Transmission in Hispanic and Low-income Preschoolers
Acronym: BESAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Rebecca Lee, Principal Investigator, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00014151
Record Dates: First submitted 2021-07-28; First posted 2022-01-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: COVID-19 Testing; Children, Preschool; Parents; Child Development; Self-Control; Exercise; Diet, Healthy
MeSH Terms: conditions — Self-Control; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participating ECE sites (N=40) will be block randomized to receive child and family back-to-ECE testing OR child and family testing plus ECE personnel biweekly testing. Of this same group of sites, half will be block randomized to complete an outdoor learning garden condition (SAGE) and have will receive waitlist. Waitlist sites will receive the garden condition delayed by one year.
Masking Description: As this is community engaged research, full transparency is required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CHILD testing (Experimental): One child and parent dyad will be tested for COVID-19 using the ASU saliva test as part of back-to-ECE safely programming. All sites will receive this condition.
  Interventions: Behavioral: CHILD back-to-ECE COVID-19 saliva testing
- CHILD+ personnel testing (Experimental): This arm receives the CHILD condition plus ECE site personnel are screened biweekly for COVID-19 using the ASU saliva test.
  Interventions: Behavioral: CHILD back-to-ECE COVID-19 saliva testing; Behavioral: ECE personnel back-to-ECE COVID-19 saliva screening
- SAGE garden (Experimental): The SAGE arm is a garden-based curriculum that emphasizes outdoor learning opportunities such as active games, songs, and garden-activities. About half of the original 40 sites (roughly evenly divided by CHILD and CHILD+) will receive this in year one, and the remaining sites will receive this condition in year two.
  Interventions: Behavioral: CHILD back-to-ECE COVID-19 saliva testing; Behavioral: ECE personnel back-to-ECE COVID-19 saliva screening; Behavioral: SAGE garden programming
- Wait list (Sham Comparator): Those in the wait list condition will receive SAGE in year two.
  Interventions: Behavioral: CHILD back-to-ECE COVID-19 saliva testing; Behavioral: ECE personnel back-to-ECE COVID-19 saliva screening

INTERVENTIONS:
Behavioral: CHILD back-to-ECE COVID-19 saliva testing — Preschool children and their parent will complete saliva COVID-19 tests at the start of the school year and after winter break as part of a back-to-ECE safely intervention. Tests may be completed during pick up, at drop off, or during school, depending on local on-campus regulations.
Behavioral: ECE personnel back-to-ECE COVID-19 saliva screening — ECE personnel will complete saliva COVID-19 tests biweekly through the school year as part of a back-to-ECE safely intervention. Tests may be completed on the ECE campus or in the parking lot, depending on local on-campus regulations
  Arms: CHILD+ personnel testing; SAGE garden; Wait list
Behavioral: SAGE garden programming — The SAGE garden programming includes installation of a garden; teacher training via Zoom and/or short videos, a binder and website support along with other accompanying materials and teacher technical support (email, text, phone); gardening supplies and gear (e.g., hats, watering cans, gloves); and delivers active songs, games, science experiments and other outdoor learning opportunities.
  Arms: SAGE garden

SUMMARY:
This study aims to get children safely back to school by (1) Child and Family Testing, (2) ECE Personnel Testing, and (3) Outdoor Learning via Garden Education.

DETAILED DESCRIPTION:
This study aims to get children safely back to school with a three strategy approach.

1. Child and Family Testing. Investigators will determine acceptability, feasibility, efficacy and scalability of testing children and families as a pre-screening strategy for re-entry to 40 CACFP-eligible ECE sites for fall 2021. Our trained bilingual ASU team (vaccinated staff and nursing students) will provide onsite testing ECE sites. Investigators will assess acceptability and feasibility via brief parent surveys and developmentally appropriate icon ratings for children, and assess efficacy as the proportion of viable samples obtained, coaching time needed to obtain one sample, and proportion of successfully obtained samples. Investigators will document costs of delivering the screening strategy (e.g., personnel, time, materials) to determine scalability. For participants testing positive for COVID-19, community health workers from Equality Health Services will provide follow-up care.
2. ECE Personnel Testing. Investigators will determine the acceptability, feasibility, efficacy and scalability of routine ECE screening of ECE personnel (teachers and aides) who have direct contact with children. Investigators will determine the acceptability of screening by 6-8 focus groups with teachers (N=80) from the 40 ECE sites above in July. Investigators will measure feasibility and efficacy (agree to test, proportion of viable samples obtained) of bi-weekly ECE site-based testing with school personnel from half (20) of the sites for fall 2021. Investigators will survey teachers to determine how acceptability toward testing relates to importance for back to ECE safety changes as vaccine uptake increases and vaccine hesitancy decreases over time. Investigators will record costs (e.g., personnel, time, materials) to determine scalability. Investigators will determine the additive efficacy of both child testing (see #1) and ECE personnel testing on attendance and enrollment. For participants testing positive for COVID-19, community health workers from Equality Health Services will provide follow-up care.
3. Outdoor Learning via Garden Education. Investigators will determine the efficacy of enhanced outdoor learning opportunities for closing the gap from the lack of in person based ECE on motor development and eating in the absence of hunger in 4 and 5 year olds. Investigators will randomize participating sites to engage in an adapted Sustainability via Active Garden Education (SAGE) garden curriculum in Spring of 2022 or wait list. Wait list sites will receive the garden and curriculum in Fall 2022. Investigators will install or enhance existing gardens in ECE sites to promote outdoor learning opportunities linked to NAEYC guidelines, and expect children in those sites to gain more rapid improvements following the learning gap. Using established protocols Investigators will test children on motor behavior and eating in the absence of hunger in Fall of 2021 (T1, baseline), prior to implementing SAGE, in Spring 2022, following SAGE implementation, and then a follow up in Fall of 2022 to determine ongoing effects.

ELIGIBILITY:
Inclusion

* Adult parents and their minor children (age 3-5)
* Children and their parents who are attending eligible early care and education (ECE) sites
* ECE site personnel (adults 18 and older) with direct contact of children attending ECE sites.

Exclusion

-Children with health-compromising conditions (e.g., food allergies) that study activities might aggravate.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1356 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Viable sample | Within six weeks from the start of school (varies by site and semester)
  Proportion of viable saliva samples obtained from children
Proportion of Children Attending ECE | within four weeks of the end of school (varies by site and semester)
  Aggregated weekly attendance of children in ECE sites and comparison (non-participating) sites.
Progressive Aerobic Cardiovascular Endurance Run (PACER) | Baseline pre-intervention
  Product-based quantitative, locomotor skills test
Progressive Aerobic Cardiovascular Endurance Run (PACER) | Post-test up to four weeks after intervention
  Product-based quantitative, locomotor skills test
Children's Activity and Movement in Preschool Study (CHAMPS) motor skill protocol | Baseline pre-intervention
  Process-based quantitative, locomotor skills test that tests skills of running, broad jumping, sliding, galloping, leaping, and hopping
Children's Activity and Movement in Preschool Study (CHAMPS) motor skill protocol | Posttest up to four week post-intervention
  Process-based quantitative, locomotor skills test that tests skills of running, broad jumping, sliding, galloping, leaping, and hopping
Eating in the absence of hunger | Baseline pre-intervention
  Behavioral, quantitative test of eating when one is not hungry
Eating in the absence of hunger | Posttest up to four weeks post-intervention
  Behavioral, quantitative test of eating when one is not hungry

SECONDARY OUTCOMES:
Acceptability and feasibility of saliva COVID-19 test | At time of COVID-19 test within six weeks from the start of school (varies by site and semester)
  Self-report survey scale that measures difficulty, satisfaction and repeatability of COVID-19 test.
Cost to obtain a sample | Time 1 at the time of COVID-19 test, Within six weeks from the start of school (varies by site and semester)
  Cost including personnel, time, materials, space to obtain a sample
Parent reports of COVID-19 household incidence | Approximately once per month following time 1, up to 10 months following time 1 (varies by site and semester)
  Brief questionnaire that measures self-report of COVID-19 cases in households enrolled in the project completed by parents approximately once per month

OTHER OUTCOMES:
Demographics | Time 1 Baseline start of the semester
  Tier 1 Common Data Element (PhenX Toolkit): Age (Demo), Annual Family Income (Demo), Employment Status (Demo), Educational Attainment (Demo), Gender (Demo), Ethnicity/Race (Demo), Health Insurance Coverage (Demo)
Vulnerability and Exposure to COVID-19 and Vaccine Acceptance | Time 1 Baseline start of the semester
  RADx-UP measure from the PhenX Toolkit of Vulnerability and Exposure to COVID-19 and Vaccine Acceptance

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Lee, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University-Downtown Campus, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data is to be shared with the RADx-UP CDCC per the DTA.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available through the RADx-UP CDCC per their governing principles.
Access Criteria: Access is through the RADx-UP CDCC.

REFERENCES:
- [Derived] Lee RE, Todd M, Oh H, Han S, Santana M, Aguilar-Troncoso J, Bruening M, Kramer JL, Leon T, Murugan V, Valdez H, Villegas-Gold M. Acceptability and Feasibility of Saliva-delivered PCR Coronavirus 2019 Tests for Young Children. Pediatrics. 2023 Jul 1;152(Suppl 1):e2022060352D. doi: 10.1542/peds.2022-060352D. PMID 37394507